CLINICAL TRIAL: NCT02840513
Title: Support by Smartphone App and Carbon Monoxide Self-monitoring for Smoking Cessation: a Randomised Controlled Trial Nested Into the Swiss HIV Cohort Study
Brief Title: Smartphone App and CO Self-monitoring for Smoking Cessation
Acronym: SMART-CO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to insufficient patient recruitment and lack of funding
Sponsor: Alain Nordmann (Other)
Responsible Party: Sponsor-Investigator, Alain Nordmann, Senior researcher, Basel Institute for Clinical Epidemiology and Biostatistics
Organization: Basel Institute for Clinical Epidemiology and Biostatistics (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AN1
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Smoking; HIV
Keywords: Smartphone app; CO self-monitoring
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone app/CO self-monitoring (Experimental): The app offers a coaching function where users receive personalized messages to encourage smoking cessation and advice for behavioural changes. For the first 4 weeks of the intervention, individuals will also be asked to blow daily into a breath carbon monoxide monitor before going to sleep. Depending on the results of the breath test, individualized messages will be delivered by the Smokelyzer feedback app to either enhance maintenance of abstinence or increase the motivation to quit. After the first 4 weeks, participants will use the breath carbon monoxide monitor at least twice a week until the end of the 6-month study. The app will react with positive feedback in individuals doing well with smoking cessation and messages to encourage individuals with difficulties quitting to smoke.
  Interventions: Other: Smartphone app/CO self-monitoring
- Control (No Intervention): Participants in the control group will be managed according to usual care as regularly provided by their SHCS physicians. Physicians will motivate patients to quit, emphasise the advantage of quitting, and provide patients with an information card that contains short advices how to quit and addresses of stop smoking clinics. The Swiss HIV Cohort Study study nurse will enter past or current use as well as of nicotine replacement therapy or use of other pharmaceutical support to quit smoking in the online study form

INTERVENTIONS:
Other: Smartphone app/CO self-monitoring — Smartphone app and carbon monoxide self-monitoring (personal device)
  Arms: Smartphone app/CO self-monitoring

SUMMARY:
This randomized controlled trial is going to evaluate whether an intervention consisting of a smartphone application to assist smokers living with HIV to quit in combination with CO self-monitoring compared to stop smoking counselling by physicians during usual care results in higher self-reported and biochemically verified smoking cessation rates at 6 months.

.

ELIGIBILITY:
Inclusion Criteria:

HIV-infected smokers ≥ 16 years and smoking ≥ 3 cigarettes /day enrolled into the Swiss HIV Cohort Study Willingness to quit smoking Speaking one or more of offical Swiss national languages or English Users of smartphone (specifically iPhone 5, 5c, 5s, 6, 6+ running iOS Version 8.0+; smartphones with resolution of at least 800x400 pixels running, Android Version 5.0+, and Android smartwatches) Informed consent

Exclusion Criteria:

Limitations in hearing, comprehension or vision problems that preclude full study participation Participants with a life expectancy of less than 12 months due to any serious medical condition

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Self-reported abstinence biochemically verified by a carbon monoxide test in-person | 6 months

SECONDARY OUTCOMES:
Differences in the number of daily cigarettes smoked from baseline to 6-month follow-up and point prevalence of abstinence (ie, no smoking in the past 7 days) at 6-month follow-up. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mdege ND, Shah S, Dogar O, Pool ER, Weatherburn P, Siddiqi K, Zyambo C, Livingstone-Banks J. Interventions for tobacco use cessation in people living with HIV. Cochrane Database Syst Rev. 2024 Aug 5;8(8):CD011120. doi: 10.1002/14651858.CD011120.pub3. PMID 39101506